CLINICAL TRIAL: NCT00301470
Title: Interest of MR Urography in the Evaluation of Functional Consequences of Urinary Tract in Children and Adults
Brief Title: Functional MR Urography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Philippe Boulangé, Directeur de la Recherche et de l'Innovation, Direction de la Recherche et de l'Innovation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI 2005 - 01
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2006-10

CONDITIONS: Ureteral Obstruction
Keywords: Ureter, obstruction; Diagnostic techniques, urological; MRI, functional
MeSH Terms: conditions — Ureteral Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MR urography — undergoing both renal scintigraphy and MR within a month

SUMMARY:
The objective of functional Uro MR is to add to an initial morphological phase, based on T2 and T1 weighted MR sequences, a sequential contrast-enhanced acquisition allowing to obtain functional semi-quantitative parameters from time-intensity curves from ROIs placed on the aorta, renal parenchyma and cavities. If the equivalence with the renal scintigraphy is demonstrated, it would be possible to have both the morphological and functional approach of an obstructed kidney in one MR examination, without exposure to diagnostic irradiation.

DETAILED DESCRIPTION:
The initial management and the follow-up of a patient presenting with chronic or intermittent obstruction is depending on clinical, biological factors and of imaging data, including the presence and degree of dilatation of pelvo-caliceal cavities and of functional consequences of such an obstruction.

The primary objectives of the study are:

* to evaluate the feasibility and reliability of the measurement of the relative renal function by MR urography compared to renal scintigraphy in the management of patients presenting with chronic and intermittent urinary obstruction in adults and children.
* if the accuracy of the two methods is demonstrated as equivalent, to conduct a medico-economic evaluation of functional MR Urography compared to renal scintigraphy, and show potential lower costs.

The secondary objectives are:

* to compare the diagnostic accuracy of various parameters of analysis of functional MR urography data, previously published in the literature, and determine indicators for predicting urinary obstruction
* to evaluate the interest of these indicators after surgical treatment of obstruction, or during the follow-up of patients
* to draw up a program of analysis and treatment of MR urography data, available for all centres whatever their MR unit.

The current study has a multicentric, observational, prospective design for the evaluation of a diagnostic strategy. It includes 16 French hospitals.

The main clinical hypothesis is that during one single MR examination, by the association of a morphological diagnostic phase and a functional phase, it will be possible to extract functional parameters having the same accuracy that renal scintigraphy in the determination of relative renal function.

The targeted recruitment is of 550 patients for two years. The MR and scintigraphy collected data will be reviewed in one site by experts at the end of the study. The university hospital of Nancy is in charge of coordinating the study.

Points of expected impact of the study are:

1. a shortening of the duration of patients management by replacing two examinations (MR and scintigraphy) by one single examination (MR )
2. a reduction of delivered exposure to diagnostic radiation, by eliminating renal scintigraphy in the initial diagnostic and follow-up of children an adults.
3. potential applications in improving the spatial resolution of MR urography after correction of artefacts such as respiratory motion.
4. the publication of clinical recommendations by the National Scientific Societies supporting the trial.

ELIGIBILITY:
Inclusion Criteria:

children (age > 1 month) and adults chronic or intermittent urinary obstruction suspected by the demonstration of uni- or bilateral dilatation of pelvo-caliceal cavities by ultrasound or CT scan.

undergoing both renal scintigraphy and MR within a month

Exclusion Criteria:

acute urinary obstruction unilateral renal agenesia and ectopic kidney renal transplantation contra-indications to MR : pace-maker, claustrophobia contra-indications to the administration of Gadolinium chelates, including pregnancy, allergy

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Main medical criterion
percentage of relative renal function of the obstructed kidney
Main economical criterion
reduction of patient's management cost in the case of a suspicion of chronic or intermittent urinary obstruction

SECONDARY OUTCOMES:
acceptability of the method by patient
reliability of the functional indicators provided by the software programme

CONTACTS AND LOCATIONS:
Overall Officials: Michel CLAUDON, PhD, Principal Investigator — Service de Radiologie
Locations (16):
- France (16):
  - Chu Angers, Angers
  - Chu Bordeaux, Bordeaux
  - Chru Lille, Lille
  - Ap-Hm Marseille, Marseille
  - Fondation LENVAL, Nice
  - AP-HP Trousseau, Paris
  - AP-HP Saint Vincent de Paul, Paris
  - AP-HP Robert Debré, Paris
  - AP-HP Bicêtre, Paris
  - Chu Poitiers, Poitiers
  - Chu Reims, Reims
  - Chu Rennes, Rennes
  - Chu Rouen, Rouen
  - Chu Strasbourg, Strasbourg
  - Chu Tours, Tours
  - CHU NANCY Hôpital Brabois enfant, Vandœuvre-lès-Nancy